CLINICAL TRIAL: NCT00199628
Title: Research Network for Neonatal Diseases Induced by Tissular Fetomaternal Alloimmunization
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I05001
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2005-09

CONDITIONS: Glomerulonephritis, Membranous; Neonatal Diseases and Abnormalities; Hemochromatosis
Keywords: fetomaternal tissular alloimmunization; Mothers having a child suffering from:; neonatal membranous glomerulonephritis; unexplained neonatal tubular defect; unexplained thrombotic microangiopathy; neonatal hemochromatosis
MeSH Terms: conditions — Glomerulonephritis, Membranous; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Hemochromatosis; Neonatal hemochromatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Problems of compatibility between a mother and her child are frequent. The most well-known case can be illustrated by the fetomaternal blood group incompatibility (rhesus factor) which can induce severe anemia of the fetus.

The investigators recently proved that incompatibility between mother and child can concern an organ leading to a tissular alloimmunization. For example, neonatal membranous glomerulonephritis (a kidney disease) can result from this mechanism.

The purpose of this network is to detect and study neonatal diseases induced by tissular fetomaternal alloimmunization. The detection of these diseases will be performed by the mother's serum analysis.

ELIGIBILITY:
Inclusion Criteria:

Mothers having a child suffering from:

* Neonatal membranous glomerulonephritis
* Unexplained neonatal tubular defect
* Unexplained thrombotic microangiopathy
* Neonatal hemochromatosis

Exclusion Criteria:

* Any cause explaining the child's disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant woman
Study Population: pregnant woman
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Guigonis, MD, Principal Investigator — Department of Pediatrics, Limoges University Hospital
Locations (1):
- Limoges University Hospital, Limoges, France